CLINICAL TRIAL: NCT02636829
Title: Validation of Self-administered Questionnaire Specifically for Assessing Calcium Intake (QALCIMUM®) in Patients With Multiple Sclerosis (MS) or Chronic Inflammatory Arthritis
Brief Title: Validation of Self-administered Questionnaire for Assessing Calcium Intake in Patients With Multiple Sclerosis or Chronic Inflammatory Arthritis
Acronym: QALCIMUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2015/ET-01; 2015-A01033-46 (Other: RCB number)
Record Dates: First submitted 2015-11-17; First posted 2015-12-22 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Sclerosis; Rheumatoid Arthritis
MeSH Terms: conditions — Multiple Sclerosis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multiple Sclerosis patients (Experimental): Patients (Multiple Sclerosis, Rheumatoid Arthritis) will be recruited during specialized consultations or hospital admissions for monitoring their chronic disease at the University Hospital of Nimes and will be divided into two distinct groups.
  Intervention: QALCIMUM questionnaire
  Intervention: Determination of calcium intake by a dietician interview
  Interventions: Other: QALCIMUM questionnaire; Other: Determination of calcium intake by a dietician interview
- Rheumatoid Arthritis patients (Experimental): Patients (Multiple Sclerosis, Rheumatoid Arthritis) will be recruited during specialized consultations or hospital admissions for monitoring their chronic disease at the University Hospital of Nimes and will be divided into two distinct groups.
  Intervention: QALCIMUM questionnaire
  Intervention: Determination of calcium intake by a dietician interview
  Interventions: Other: QALCIMUM questionnaire; Other: Determination of calcium intake by a dietician interview

INTERVENTIONS:
Other: QALCIMUM questionnaire — All patients will fill out the QALCIMUM questionnaire.
Other: Determination of calcium intake by a dietician interview — All patients will have an interview with a dietician who performs a food survey serving as a reference (gold standard) and based on data from CIQUAL *.
  * CIQUAL Data: Nutritional food composition table available on the website of the ANSES (National Agency for Sanitary Security of Food, Environment and Labour), published by the Observatory of the Nutritional Quality of Foods. This table includes 1500 sheets of 58 nutritional components. The data is integrated into the software (DATAMEAL) for calculating the ingesta parameters at the Nîmes University Hospital.

SUMMARY:
The main objective of this study is to measure, in patients with MS or Chronic Inflammatory Arthritis (CIA), the correlation between two calcium intake assessment methods: A self assessment questionnaire of calcium intake (QALCIMUM®) versus a food survey serving as a reference (gold standard) and based on data from CIQUAL *.

* CIQUAL Data: Nutritional food composition table available on the website of the ANSES (National Agency for Sanitary Security of Food, Environment and Labour), published by the Observatory of the Nutritional Quality of Foods. This table includes 1500 sheets of 58 nutritional components. The data is integrated into the software (DATAMEAL) for calculating the ingesta parameters at the Nîmes University Hospital.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To estimate the average calcium intake and variability in a population of MS patients and the proportion of patients at risk for osteoporosis.

B. To estimate the average calcium intake and variability in a population of CIA patients and the proportion of patients at risk for osteoporosis.

C. To describe the dietary changes observed in MS or CIA patients .

D. To estimate the administration time of the QALCIMUM® self-questionnaire.

E. Estimate calcium intake means and variability in a population of patients with MS or CIA and the proportion of patients at risk of osteoporotic fracture

F. To assess the quality of life of patients with MS or CIA

G. To evaluate endogenous mean vitamin D production in a population of patients with MS or CIA

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patient with confirmed diagnosis of multiple sclerosis or chronic inflammatory arthritis (rheumatoid arthritis, spondyloarthritis, psoriatic arthritis)

Exclusion Criteria:

* The patient is participating in another biomedical research study
* The patient has participated in another biomedical research study in the past 3 months
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or under guardianship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The subject is not able to complete a self-administered questionnaire

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Calcium intake (mg/day) | Day 0
  As determined by a consultation with a dietician.
The QALCIMUM questionnaire | Day 0

SECONDARY OUTCOMES:
Patient diet (qualitative) | Day 0
  Patient diet classified as: normal; vegetarian, vegetalian; Seignalet; Kousmine; other.
QALCIMUM questionnaire administration time (minutes) | Day 0
The GRIO questionnaire | Day 0
  GRIO = Osteoporosis Research and Information Group
The FRAX questionnaire | Day 0
  FRAX = WHO Fracture RISK Assessment Tool
Quality of Life questionnaire: MSIS29 (MS Impact Scale) | Day 0
Quality of Life questionnaire: TLSQOL10 | Day 0
Quality of Life questionnaire: TLS Coping | Day 0
The Vitamin D questionnaire | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvenot, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France